CLINICAL TRIAL: NCT01971749
Title: Multicenter, Prospective, Observational Study of of Treatment of Unprotected Left Main Coronary Artery Stenosis in Andalucía
Brief Title: Register of Treatment of Unprotected Left Main Coronary Artery Stenosis in Andalucía
Acronym: RETRATO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundación Pública Andaluza Progreso y Salud (Other)
Responsible Party: Sponsor
Organization: Andalusian Network for Design and Translation of Advanced Therapies (Other)
Other Study IDs: CSG-TCI-2012-01
Record Dates: First submitted 2013-10-18; First posted 2013-10-29 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-08

CONDITIONS: Unprotected Left Main Coronary Artery Stenosis
Keywords: Coronary stent procedure (CSP; Coronary-artery bypass grafting (CABG)
MeSH Terms: interventions — Coronary Artery Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Unprotected left main coronary artery stenosis patients
  Interventions: Procedure: Coronary stent procedure (CSP); Procedure: Coronary-artery bypass grafting (CABG)

INTERVENTIONS:
Procedure: Coronary stent procedure (CSP)
Procedure: Coronary-artery bypass grafting (CABG)

SUMMARY:
Register of treatment of unprotected left main coronary artery stenosis in Andalucia (RETRATO).

ELIGIBILITY:
Inclusion Criteria:

* New diagnosed of unprotected left main coronary artery stenosis (lesion ≥50%)
* Have signed informed consent

Exclusion Criteria:

* Participating in other research protocol
* Inability to follow a monitoring

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients with unprotected left main coronary artery stenosis in Andalucia who can follow a year monitoring in participating centers
Sampling Method: Non-Probability Sample
Enrollment: 315 (Estimated)
Dates: Start 2013-05; Primary Completion 2015-12 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Measure the MACE survival in the coronary-artery bypass grafting (CABG) group and in the coronary stent procedure (CSP) group, to identify the differences between both groups in the short and medium-term follow up | 12 months
  MACE= Major Adverse Cardiac Event (e.g., acute myocardial infarction, ischaemic stroke, coronary arterial occlusion, death)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Sánchez González, Principal Investigator — Hospital Carlos Haya
Locations (6):
- Spain (6):
  - Hospital Torrecárdenas, Almería
  - Hospital Universitario San Cecilio, Granada
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Juan Ramón Jiménez, Huelva
  - Hospital Carlos Haya, Málaga
  - Hospital Clínico Universitario Virgen de la Victoria, Málaga